CLINICAL TRIAL: NCT06928636
Title: Supper Heroes: Randomized Controlled Trial to Examine the Impact of an Online Environmentally Friendly Eating Intervention for Families
Brief Title: Supper Heroes: Examining the Impact of an Online Eating Intervention for Families
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Responsible Party: Principal Investigator, Jess Haines, Professor, University of Guelph
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Supper Heroes: RCT
Record Dates: First submitted 2025-03-27; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-03

CONDITIONS: Eating Behaviors
Keywords: food waste; environmentally friendly; plant-based foods
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Other): Families randomized to the control group will receive weekly emails for 7 weeks about environmentally friendly habits.
  Interventions: Behavioral: Monthly emails about environmentally friendly habits
- Supper Heroes online environmentally friendly eating intervention for families (Experimental): Families randomized to the intervention group will complete a 7-week Supper Heroes program that includes activities focused on making more meals at home, reducing food waste, and eating more plant-based foods.
  Interventions: Behavioral: Supper Heroes online environmentally friendly eating intervention for families

INTERVENTIONS:
Behavioral: Supper Heroes online environmentally friendly eating intervention for families — Families randomized to the intervention group will complete a 7-week Supper Heroes program that includes activities focused on making more meals at home, reducing food waste, and eating more plant-based foods.
  Arms: Supper Heroes online environmentally friendly eating intervention for families
Behavioral: Monthly emails about environmentally friendly habits — Families randomized to the control group will receive monthly emails for 6 months about environmentally friendly habits.
  Arms: Control Group

SUMMARY:
This study will examine the effectiveness of the online family-based program focused on sustainable eating compared to weekly emails about environmentally friendly behaviours.

DETAILED DESCRIPTION:
The investigators will conduct a family-level RCT following CONSORT guidelines: families will be randomly allocated into control and intervention groups. The control group will receive an email once a week for 7 weeks with information about environmentally friendly habits.

The intervention group will participate in the 7-week online Supper Heroes program consisting of 7 online "missions" completed over 7 weeks. Each mission includes tasks for families to complete, including reading infographics, watching short videos, participating in family-based activities, and sharing their progress. Parents will receive 2 text messages each week with information about the program. Families will also receive a toolkit to support their participation which will contain cookbooks, a potato brush, grocery planning tools, and a note that orients them to what is included. It will take approximately 1-2 hours per mission to complete all activities.

* Infographics: Each mission will contain brief, 1-2-page infographics for families to read. Topics are related to the mission theme for that week. For example, families may learn about tips for grocery shopping and meal planning as well as information about plant-based proteins.
* Videos: Similar to the infographics, short, 1-5-minute online videos will be related to the theme of the mission participants are completing. For example, families will watch a short, animated video about grocery shopping.
* Family-based activities: During each mission, participants will be invited to participate in a family-based activity such as follow-along cooking videos, doing an audit of their fridge, and creating a grocery shopping list.
* Sharing: Families will be asked to share their experiences for each mission on an online community share board by providing a photo and/or text.

ELIGIBILITY:
Inclusion Criteria:

* have at least one child 9-12 years old
* live in Ontario, Canada
* have access to the internet
* can respond to English surveys

Exclusion Criteria:

* parent(s) with prior nutrition and food education (e.g., degree in nutrition, culinary arts training)
* families with food allergies that would prevent them from participating in the intervention (e.g., soy products, beans or lentils)
* families who are vegetarian or vegan

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Decrease in avoidable food waste | 15 months
  The amount of avoidable food waste generated is measured as the difference in weight (grams) between baseline (T0), post-intervention/control (T1), and 6-month follow-up (T2), as assessed by weighed food waste diaries. Participants will complete a food waste diary using a provided kitchen scale and detailed instructions on how to do so. The amount of avoidable food waste will be compared between participants in the Supper Heroes intervention group and those in the control group.
  Measurement Tool: Food waste diary and kitchen scale.
  Unit of Measure: Families will be asked to list all food thrown away, the weight of the food (gams) and the reason the food was thrown away (e.g., it went bad) for 7 days.
  Time Points: Baseline (T0): post-intervention/control (T1 - after completion of either intervention or control activities, 7 weeks); follow-up (T2 - 6 months after completing the intervention or control activities).

SECONDARY OUTCOMES:
Increased intake of plant-based foods among parents and children. | 15 months
  The amount of plant-based foods consumed by parents and children is measured as the mean servings of plant-based foods, as assessed by a web-based food frequency questionnaire. This will be compared between participants in the Supper Heroes intervention group and those in the control group.
  Measurement Tool: Food frequency questionnaire adapted from Canadian Diet History Questionnaire II (National Cancer Institute, n.d.)
  Unit of Measure: Servings of plant-based foods consumed per day
  Time Points: Baseline (T0): post-intervention/control (T1 - after completion of either intervention or control activities, 7 weeks); follow-up (T2 - 6 months after completing the intervention or control activities).
  National Cancer Institute. (n.d.). Diet History Questionnaire (DHQ2). U.S. Department of Health and Human Services. Retrieved April 3, 2025, from https://epi.grants.cancer.gov/dhq2/
Decreased intake of red and processed meats among parents and children. | 15 months
  The amount of red and processed meats consumed by parents and children, measured as the average daily intake (servings) of red and processed meats, as assessed by a web-based food frequency questionnaire. This will be compared between participants in the Supper Heroes intervention group and those in the control group.
  Measurement Tool: Food frequency questionnaire adapted from Canadian Diet History Questionnaire II (National Cancer Institute, n.d.)
  Unit of Measure: Servings of red and processed meats consumed per day
  Time Points: Baseline (T0): post-intervention/control (T1 - after completion of either intervention or control activities, 7 weeks); follow-up (T2 - 6 months after completing the intervention or control activities).
  National Cancer Institute. (n.d.). Diet History Questionnaire (DHQ2). U.S. Department of Health and Human Services. Retrieved April 3, 2025, from https://epi.grants.cancer.gov/dhq2/

OTHER OUTCOMES:
Evaluate mechanisms of behaviour change. | 15 months
  The changes in parents' and children's attitudes, subjective norms, and perceived behavioral control, measured using items previously validated in the feasibility study (Eckert et al., 2025), as potential mediators of the intervention effects on the primary and secondary outcomes. These constructs will be assessed before and after the intervention to determine their role in mediating changes in behavior, such as the intake of plant-based foods and red/processed meats.
  Time Points: Baseline (T0): post-intervention/control (T1 - after completion of either intervention or control activities, 7 weeks).
  Eckert KF, Agostinelli J, Laila A, Alexander C, Parizeau K, von Massow M, Duncan AM, Hesketh KD, Ma DWL, Haines J. Feasibility, acceptability, and preliminary impact of "Supper Heroes", a family-based sustainable diet intervention. Appetite. 2025 Feb 1;206:107849. doi: 10.1016/j.appet.2025.107849. Epub 2025 Jan 7. PMID: 39788349.

CONTACTS AND LOCATIONS:
Overall Officials: Jess Haines, PhD, Principal Investigator — University of Guelph
Locations (1):
- University of Guelph, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No